CLINICAL TRIAL: NCT05215210
Title: The Effect of Long-term Momordica Charantia Supplementation on Blood Glucose Levels
Acronym: Bitter-Zoet 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wageningen University and Research (Other)
Responsible Party: Principal Investigator, Diederik Esser, Project leader clinical trials, Wageningen University and Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NL79294.091.21
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Glucose, High Blood; Impaired Glucose Tolerance
Keywords: bitter gourd; pre-diabetes; fasting blood glucose
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Supplements will be labeled A and B by a scientist who is not involved in this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bitter-gourd (Experimental): dried bitter-gourd supplements
  Interventions: Other: Bitter-gourd
- Cucumber (Active Comparator): dried cucumber supplements
  Interventions: Other: Cucumber

INTERVENTIONS:
Other: Bitter-gourd — 12-week intervention of 3.6 grams of dried bitter-gourd supplements
  Arms: Bitter-gourd
Other: Cucumber — 12-week intervention of 3.6 grams of cucumber supplements
  Arms: Cucumber

SUMMARY:
The study is a parallel, double blind, controlled trial in which study participants will receive a 12-week intervention with 3.6 g/d dried bitter-gourd supplements or a reference intervention with 3.6 g/d dried cucumber supplements. Research subjects will come to the research facility for a test day on four occasions, with an interval of 4 weeks. The main study parameter is fasting levels of plasma glucose.

DETAILED DESCRIPTION:
Bitter gourd (BG) (Momordica charantia) is a highly nutritive vegetable from the cucumber family. The objective is to assess the impact of 12-weeks of BG supplementation on blood glucose levels in subjects with impaired fasting glucose levels. In a previous trial (Bitter-Zoet NL70259.081.19) the short-term effects of BG (4 weeks) were studied, but no effect was observed. In the current trial a different BG cultivar is chosen, the intervention period is prolonged, the dosage per day is higher and study subjects with slightly higher fasting blood glucose levels will be included. The study is a parallel, double blind, controlled trial in which study participants will receive a 12-week intervention with 3.6 g/d dried bitter-gourd supplements or a reference intervention with 3.6 g/d dried cucumber supplements. Research subjects will come to the research facility for a test day on four occasions, with an interval of 4 weeks. The main study parameter is fasting levels of plasma glucose. Secondary outcome measures are glucose tolerance, HbA1c, insulin and HOMA-IR and HOMA-B levels.

ELIGIBILITY:
Inclusion Criteria:

* age 40-75yrs
* BMI >25 kg/m2
* Having a fasting glucose >6.1 mmol/L

Exclusion Criteria:

* Use of medication/supplements that may influence the study results, such as metformin, gliclazide, glimepiride, tolbutamide, insulin, sitagliptin (DPP4 inhibitor), liraglutide (GLP-1 agonist), acarbose, repaglinide, pioglitazone, corticosteroids (systemically) , SGLT-2 inhibitors, (judged by our research physician)
* Having a fasting glucose >11.0 mmol/L
* History of gastro-intestinal surgery or having (serious) gastro-intestinal complaints
* History of liver dysfunction (cirrhosis, hepatitis) or liver surgery
* Reported slimming, medically prescribed or other extreme diets
* Reported weight loss or weight gain of > 5 kg in the month prior to pre-study screening
* Not willing to give up blood donation during the study
* Current smokers
* Alcohol intake ≥14 glasses (women) or >21 glasses (men) of alcoholic beverages per week, on average
* pregnant or lactating (self-reported)
* Abuse of illicit drugs (soft- and hard drugs)
* Food allergies for products that we use in the study
* Participation in another clinical trial at the same time
* Being an employee of the Food, Health & Consumer Research group of Wageningen Food & Biobased Research or dept. human nutrition and health of Wageningen University.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-03-23 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
change in fasting plasma glucose concentrations | Baseline (before supplementation (T0)), after 4 weeks (T2), 8 weeks (T3) and 12 weeks (T4)
  marker for glucose metabolism

SECONDARY OUTCOMES:
change in 2hour plasma glucose concentrations after a 75-gram OGTT | Baseline (before supplementation (T0)) and after 12 weeks (T4)
  marker for glucose metabolism
change in HbA1c | Baseline (before supplementation (T0)), after 4 weeks (T2), 8 weeks (T3) and 12 weeks (T4)
  marker for glucose metabolism
change in insulin | Baseline (before supplementation (T0)), after 4 weeks (T2), 8 weeks (T3) and 12 weeks (T4)
  marker for glucose metabolism
change in HOMA-IR levels | Baseline (before supplementation (T0)), after 4 weeks (T2), 8 weeks (T3) and 12 weeks (T4)
  marker for glucose metabolism
change in HOMA-B levels | Baseline (before supplementation (T0)), after 4 weeks (T2), 8 weeks (T3) and 12 weeks (T4)
  marker for glucose metabolism

OTHER OUTCOMES:
change in ALAT | Baseline (before supplementation (T0)), after 4 weeks (T2), 8 weeks (T3) and 12 weeks (T4)
  liver enzyme (study safety parameter)
change in ASAT | Baseline (before supplementation (T0)), after 4 weeks (T2), 8 weeks (T3) and 12 weeks (T4)
  liver enzyme (study safety parameter)
change in eGFR | Baseline (before supplementation (T0)), after 4 weeks (T2), 8 weeks (T3) and 12 weeks (T4)
  estimated glomerular filtration rate (study safety parameter)
change in creatinine | Baseline (before supplementation (T0)), after 4 weeks (T2), 8 weeks (T3) and 12 weeks (T4)
  kidney function (study safety parameter)

CONTACTS AND LOCATIONS:
Overall Officials: Sandra van der Haar, MSc, Principal Investigator — Stichting Wageningen Research
Locations (1):
- Stichting Wageningen Research, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No